CLINICAL TRIAL: NCT00768976
Title: Study of Patient Satisfaction With the Cancer Clinical Trial Experience
Status: Completed | Type: Observational
Sponsor: Summa Health System (Other)
Responsible Party: Principal Investigator, Joyce Neading, Program Director, Cancer Research & Cancer Registry, Summa Health System
Other Study IDs: Clinical trial experience
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Cancer
Keywords: Participant must have participated in a clinical trial conducted by the Summa Health System Hospitals Cancer Research Program.; Participant should have been registered for clinical trial participation three months prior to receiving the satisfaction survey.
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to evaluate the quality of the clinical trial experience of cancer patients participating in cancer research studies through Summa Health System Hospitals Cancer Research Program by evaluating patient satisfaction regarding reasons for participating, facility, consent and treatment, personal issues and overall assessment.

The secondary objective of this study is to determine areas for improvement to make the patient's clinical trial experience a satisfying and positive journey.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have participated in a clinical trial conducted by the Summa Health System Hospitals Cancer Research Program.
* Participant should have been registered for clinical trial participation three months prior to receiving the satisfaction survey.

Exclusion Criteria:

* Participant has withdrawn consent for clinical trial participation and/or follow up.
* Participant has a major medical illness that would prevent completion of the survey.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant must have participated in a clinical trial conducted by the Summa Health System Hospitals Cancer Research Program.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of surveys to determine if there are opportunities for performance and/or quality improvement projects.patient satisfaction regarding reasons for participating, facility, consent and treatment, personal issues and overall assessment. | Survey will be sent to subject 3 months after study registration

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Neading, RHIT, CTR, Principal Investigator — Summa Health System